CLINICAL TRIAL: NCT06216977
Title: CODA-POP Surgery: Clears On the Day of Anesthesia Permissible up to One-Hour Prior to Surgery - A Prospective Randomized and Blind Trial
Brief Title: Clears On the Day of Anesthesia Permissible up to One-Hour Prior (CODA-POP) to Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI passed away
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, yafen liang, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-23-0868
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Nutrition
Keywords: Nil Per Os (NPO); stomach volume; gastric volume; Aspiration
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear Liquids Arm (Experimental)
  Interventions: Other: Clear Liquids
- Standard Of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Clear Liquids — Participants will not take anything by mouth after midnight the day before surgery but will be given 12 ounce clear liquid (Sugar-free Gatorade) at bedside at the pre-operative holding area
  Arms: Clear Liquids Arm
Other: Standard of Care — Participants will not take anything my mouth after midnight day before surgery
  Arms: Standard Of Care

SUMMARY:
The purpose of this study is to assess whether residual gastric volumes in patients who receive clear liquids one hour prior to time of procedure is non-inferior compared to patients who are NPO past midnight, to compare efficiency and flexibility of operating room scheduling between two fasting conditions, to assess patient satisfaction and post-operative nausea, vomiting, pain, hunger and thirst.

and to assess wound healing and post-operative complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing laparoscopic cholecystectomy during the day or night of a weekday (including those consented on a Friday who get postponed to a weekend surgery start time).
* Modified rapid sequence intubation (mRSI)

Exclusion Criteria:

* History of reflux disease
* History of hiatal hernia
* History of esophageal disease
* History of gastroparesis
* Known history of difficult airway or planned fiberoptic intubation
* HbA1c greater than 12
* Pregnant women
* Prisoner
* Procedures conducted on weekends and holidays
* Emergency or non-elective procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Residual Gastric Volume in mL/kg | At time of intubation (about 1 hour after fluid intake)

SECONDARY OUTCOMES:
Number of participants with observed emesis | During perioperative period which includes preoperative, intraoperative and post operative time (about 4 hours)
Number of participants with subjective pre-operative nausea | at baseline
Number of participants with subjective post-operative nausea | within 24 hours of surgery
Number of participants with production of oropharyngeal secretions | During the perioperative period which includes preoperative, intraoperative and post operative time (about 4 hours)
Number of participants with wound dehiscence | postoperative follow up appointment (about 1 month after surgery)
Number of participants with intraoperative complications | From start of surgery to end of surgery
Amount of post-operative pain medications needed | at first clinic appointment (about 1 month after surgery)
Overall patient satisfaction as assessed by the Press-Ganey Questionnaire | within 48-96 hours of surgery
  This is a 10 item questionnaire and each is scored from 1(very poor) to 5(very good) , maximum score of 50 a higher number indicating better outcome

CONTACTS AND LOCATIONS:
Overall Officials: George Williams, MD, FASA, FCCM, FCCP, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No